CLINICAL TRIAL: NCT03702257
Title: Intérêt Diagnostique et Pronostique de la présence d'Anticorps spécifiques du Donneur Intra-greffon Dans le Rejet Humoral en Transplantation Pulmonaire
Brief Title: DSA Intragraft in Lung Transplantation: Diagnostic and Prognostic Value in Antibody Mediated Rejection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7039
Record Dates: First submitted 2018-10-08; First posted 2018-10-11 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Lung Transplant Recipient; Donor Specific Antibodies; Antibody Mediated Rejection
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bronchial fibroscopy (Other): Bronchial fibroscopy with trans-bronchial biopsies
  Interventions: Procedure: bronchoscopy.

INTERVENTIONS:
Procedure: bronchoscopy. — gDSAs are studied on cryopreserved biopsies obtained during bronchoscopy. The technique is the one described by Visentin J.

SUMMARY:
The diagnosis of AMR in lung transplant recipients is difficult and often comes too late, because of lack of standardized definition. The diagnosis is nowadays based on an expert multidisciplinary approach involving clinical, histopathological and immunological criteria.

Hypothesis: the presence of intragraft donor specific antibodies (gDSAs) could be used as a new diagnostic tool for AMR in lung transplant recipients Study Objectives: to evaluate, in lung transplant patients with circulating DSAs, the diagnostic value of gDSAs in AMR and to analyze its prognostic value on graft outcome.

ELIGIBILITY:
Inclusion criteria:

* Patient older than 18 years
* Transplanted pulmonary or cardiopulmonary patient
* And developing circulating anti-HLA antibodies directed against the graft or "DSA" at a threshold > 1000 of MFI in the 30 days preceding the inclusion visit
* Affiliation to the French social security
* Patient able to understand the objectives and risks related to research and to give informed, dated and signed consent

Exclusion criteria:

* Patient whose anti-HLA antibodies are not directed against the graft (no DSA)
* Contraindication to performing a bronchial fibroscopy with transbronchial biopsies
* Treatment with intravenous immunoglobulin (less than 1 month before inclusion) or Rituximab (less than 6 months before inclusion)
* Plasma exchanges (less than 3 months before inclusion)
* Risk of bleeding predictable (crushing disorder, impossibility of stopping the offending treatments)
* Impossibility of giving the subject informed information
* Subject under the protection of justice Subject under guardianship or curatorship
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of AMR | 2 years
  Sensitivity and specificity of the presence of gDSA for the diagnosis of AMR in lung transplant recipients with circulating DSA, as established by an expert pathologist panel and in accordance with recent international recommendations

SECONDARY OUTCOMES:
Comparaison in gDSA+ vs gDSAs- patients | 2 years
  Incidence of graft loss

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hôpital Marie Lannelongue, Le Plessis-Robinson
  - CHU Nord, Marseille
  - Hôpital Bichat, Paris
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: Undecided